CLINICAL TRIAL: NCT01844219
Title: Accuracy of Pre-existing Risk Scoring Models for Predicting Acute Kidney Injury in Patients Who Underwent Aortic Surgery Using a Gray Zone Approach
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jong Hwan Lee, Assistant Professor, Samsung Medical Center
Other Study IDs: 2013-03-059-001
Record Dates: First submitted 2013-04-28; First posted 2013-05-01 (Estimated); Last update posted 2013-12-25 (Estimated); Status verified 2013-12

CONDITIONS: Aortic Surgery; Postoperative Acute Kidney Injury
Keywords: aortic surgery; acute kidney injury; gray zone approach
MeSH Terms: conditions — Acute Kidney Injury | interventions — Elective Surgical Procedures; Clonal Hematopoiesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients who underwent aortic surgery: Patients who underwent aortic surgery in Samsung Medical Center during the period between 2004 and 2010
  Interventions: Procedure: elective or emergency aortic surgery (including ascending, arch, descending thoracic aorta)

INTERVENTIONS:
Procedure: elective or emergency aortic surgery (including ascending, arch, descending thoracic aorta)
  Other Names: graft interposition of thoracic aorta

SUMMARY:
Acute kidney injury after cardiac surgery has been reported to increase morbidity and mortality. Several risk scoring models for prediction of aortic kidney injury after cardiac surgery have been developed. However, predictive accuracy of these models is stil unclear. The aim of this study is to evaluate the accuracy of four pre-existing prediction models using a gray zone approach in patients who underwent aortic surgery in our institution.

DETAILED DESCRIPTION:
Acute kidney injury after cardiac surgery has been reported to increase morbidity and mortality. Several risk scoring models for prediction of aortic kidney injury after cardiac surgery have been developed. However, predictive accuracy of these models is stil unclear. The aim of this study is to evaluate the accuracy of four pre-existing prediction models (AKICS, Wijeysundera, Mehta, and Thakar model)using a gray zone approach in patients who underwent aortic surgery in our institution. Based on receiver operating characteristic (ROC) curve analysis, we will construct a gray zone using the cut-off values with a sensitivity of < 90%, and a specificity of < 90% (diagnostic tolerance of 10%).

ELIGIBILITY:
Inclusion Criteria:

* Those who underwent elective or emergency aortic surgery in Samsung Medical Center during between 2004 and 2010.

Exclusion Criteria:

* missing laboratory data
* preoperative hemodialysis
* death during or within 48 hours after surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Those who underwent elective or emergency aortic surgery in Samsung Medical Center during between 2004 and 2010.
Sampling Method: Non-Probability Sample
Enrollment: 375 (Actual)
Dates: Start 2013-04; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
presence of acute kidney injury | within 48 hour after aortic surgery
  1. abrupt (within 48 hours) reduction in kidney function currently defined as
  2. absolute increase in serum creatinine of more than or equal to 0.3 mg/dl (≥ 26.4 μmol/l),
  3. a percentage increase in serum creatinine of more than or equal to 50% (1.5-fold from baseline), or
  4. a reduction in urine output (documented oliguria of less than 0.5 ml/kg per hour for more than six hours)

SECONDARY OUTCOMES:
Gray zone range of each risk scoring model | within 48 hours
  Thresholds with as a sensitivity of < 90% and a specificity of < 90%.
Number of patients in the gray zone | within 48 hours after aortic surgery
  Number of patients in the gray zone in each risk scoring model

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Sungkyunkwan University, School of Medicine, Seoul, South Korea